CLINICAL TRIAL: NCT02372786
Title: A Double Blind Randomized Controlled Trial Comparing the Efficacy of 7% Lidocaine / 7% Tetracaine Cream Versus 2,5% Lidocaine / 2,5% Prilocaine Cream for Local Anaesthesia During Laser Treatment of Acne Keloidalis Nuchae and Tattoo Removal
Brief Title: 7% Lidocaine/7% Tetracaine Cream Versus 2,5% Lidocaine / 2,5% Prilocaine Cream
Acronym: OPTICA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, M.B.A. van Doorn, MD, PhD, Erasmus Medical Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MEC-2014-517_OPTICA
Record Dates: First submitted 2015-02-12; First posted 2015-02-26 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Tattoo; Acne Keloidalis Nuchae
Keywords: 7% lidocaine / 7% tetracaine cream; 2,5% lidocaine / 2,5% prilocaine cream
MeSH Terms: conditions — Acne Keloid | interventions — Lidocaine, Prilocaine Drug Combination; Lidocaine; Lasers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acne Keloidalis Nuchae (Other): 2,5% lidocaine / 2,5% prilocaine cream and 7% lidocaine / 7% tetracaine cream will be applied for 60 minutes. After removal of the creams patients will recieve laser hair removal treatment using a neodymium-doped yttrium aluminium garnet (Nd:Yag) laser.
  Interventions: Drug: 2,5% lidocaine / 2,5% prilocaine cream; Drug: 7% lidocaine / 7% tetracaine cream; Device: Neodymium-doped yttrium aluminium garnet (Nd:Yag) laser
- Tattoo (Other): 2,5% lidocaine / 2,5% prilocaine cream and 7% lidocaine / 7% tetracaine cream will be applied for 60 minutes. After removal of the creams patients will recieve laser tattoo removal treatment using a Q-switched nd Yag laser.
  Interventions: Drug: 2,5% lidocaine / 2,5% prilocaine cream; Drug: 7% lidocaine / 7% tetracaine cream; Device: Q-switched nd Yag laser

INTERVENTIONS:
Drug: 2,5% lidocaine / 2,5% prilocaine cream — The treatment area will be divided in two equal parts with white markings. Between these two areas an area of 1 cm will be marked. This area will be left untreated, to avoid possible spill-over effects of the two anaesthetic creams. A thick layer of 2,5% lidocaine / 2,5% prilocaine cream will be applied on one side to the intact skin under plastic occlusion (average of 1,5-2g per 10 cm2) 60 minutes before laser treatment.
  Other Names: Emla®
Drug: 7% lidocaine / 7% tetracaine cream — The treatment area will be divided in two equal parts with white markings. Between these two areas an area of 1 cm will be marked. This area will be left untreated, to avoid possible spill-over effects of the two anaesthetic creams. A thin layer of 7% lidocaine / 7% tetracaine cream (1mm) will be applied on the other side to the intact skin (average of 1,3g Pliaglis per 10 cm2) 60 minutes before laser treatment.
  Other Names: Pliaglis®
Device: Neodymium-doped yttrium aluminium garnet (Nd:Yag) laser — Acne keloidalis nuchae: during this study a 1064 nm Nd:yag laser with a spot size of 7-10 mm, and a fluence of 35-60J/cm2, (depending on the effective and safe clinical response), a pulse duration of 20-35 ms and 2 passes will be used.
  Arms: Acne Keloidalis Nuchae
Device: Q-switched nd Yag laser — Tattoo removal: we will use a 3 mm spotsize and a fluence depending on the absorption of the laser light, which is visible as skin whitening.
  Arms: Tattoo

SUMMARY:
The purpose of this study is to compare the efficacy of 7% lidocaine / 7% tetracaine cream and 2,5% lidocaine / 2,5% prilocaine cream in reducing self-reported pain during a single laser procedure in the treatment of acne keloidalis nuchae and tattoo removal.

DETAILED DESCRIPTION:
In this study we will compare the efficacy of 7% lidocaine / 7% tetracaine cream and 2,5% lidocaine / 2,5% prilocaine cream in reducing self-reported pain during a single laser procedure in the treatment of acne keloidalis nuchae and tattoo removal. Patients will be asked to fill in questionnaires to:

* assess the severity of pain experienced (VAS score) during laser treatment,
* evaluate whether the pain relief is adequate and,
* evaluate the amount of money patients would be willing to pay for the cream that provided the 'best' pain relief.

One week after the visit the patient will have a telephone consultation. The patients will be asked if they experienced any symptoms, which will be recorded as adverse events.

ELIGIBILITY:
Inclusion Criteria:

* • Subject has provided written informed consent;

  * Subject is ≥ 18 years of age at time of screening;
  * Group A: subjects with acne keloidalis nuchae;
  * Group B: subjects with an uniform, black, professionally placed tattoo

Exclusion Criteria:

* • Known sensitivity to any components of the test materials;

  * Pregnant or breast-feeding women;
  * Use of any other pain medication during past 24 hours prior to the laser treatment;
  * Damaged skin at the designated treatment site;
  * Blister formation and/or scar formation after test-treatment with standard laser settings;
  * Any medical or psychiatric condition which, in the investigator's opinion, would preclude the participant from adhering to the protocol or completing the study per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Self-reported pain (10 point visual analog scale). | 5 minutes

SECONDARY OUTCOMES:
adequate pain relief (yes/no); | 10 minutes
willing to spend around 25 euro for best pain relief (yes/no). | 10 minutes
To monitor the nature and frequency of adverse events | one week

CONTACTS AND LOCATIONS:
Overall Officials: Martijn van Doorn, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands